CLINICAL TRIAL: NCT05294640
Title: Bacteriostatic Saline as a Local Anesthetic in Minor Eyelid Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-36276
Record Dates: First submitted 2022-03-08; First posted 2022-03-24 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Eyelid Tumor; Eyelid Bump; Eyelid Deformity; Eyelid Abscess; Eyelid Boil; Eyelid Papilloma; Anesthesia, Local; Ophthalmology
Keywords: Oculoplastics; Local Anesthesia; Eyelid Anesthesia; Periocular Anesthesia
MeSH Terms: conditions — Eyelid Neoplasms; Hordeolum | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patient and provider performing procedure will be masked to local anesthesia type
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bacteriostatic Saline as Local Anesthesia (Experimental): Patients receiving bacteriostatic saline as local anesthesia for in-office minor eyelid procedures at University of California, San Francisco Medical Center, Oculoplastics department
  Interventions: Drug: 0.9% Bacteriostatic Local Anesthetic Injection; Procedure: Eyelid Lesion Removal
- Lidocaine with Epinephrine as Local Anesthesia (Active Comparator): Patients receiving lidocaine with epinephrine as local anesthesia for in-office minor eyelid procedures at University of California, San Francisco Medical Center, Oculoplastics department
  Interventions: Drug: 1% Lidocaine with 1:100,000 epinephrine Local Anesthetic Injection; Procedure: Eyelid Lesion Removal

INTERVENTIONS:
Drug: 0.9% Bacteriostatic Local Anesthetic Injection — Following research and procedural consent, local anesthetic injection will be carried out using a standard 1 cc of local anesthetic corresponding to the study arm (0.9% bacteriostatic saline or 1% lidocaine with 1:100,000 epinephrine). Prior to anesthetic administration, the procedure site will be cleaned using standard measures. A 30 gauge needle on a 3 centimeter cubed volume syringe will be utilized. Five minutes will be given for local anesthetic to take effect.
  Arms: Bacteriostatic Saline as Local Anesthesia
Drug: 1% Lidocaine with 1:100,000 epinephrine Local Anesthetic Injection — Following research and procedural consent, local anesthetic injection will be carried out using a standard 1 cc of local anesthetic consisting of a commercially available mixture of 1% lidocaine with 1:100,000 epinephrine. Prior to anesthetic administration, the procedure site will be cleaned using standard measures. A 30 gauge needle on a 3 centimeter cubed volume syringe will be utilized. Five minutes will be given for local anesthetic to take effect.
  Arms: Lidocaine with Epinephrine as Local Anesthesia
Procedure: Eyelid Lesion Removal — Following anesthesia administration, patient will proceed with recommended eyelid lesion removal. The procedure site will be cleaned according to standard protocol, and standard technique for lesion removal will be performed, which will vary according to type of lesion but may involve use of Westcott scissors, forceps, #15 or #11 blades or other oculoplastics administration. The exact procedural details will be at the discretion of the surgeon.

SUMMARY:
The investigators aim to assess whether bacteriostatic saline provides the same level of anesthesia as traditional local anesthesia while reducing pain associated with medication infusion in minor eyelid procedures

DETAILED DESCRIPTION:
Benzoyl alcohol is an aromatic alcohol that has been used in healthcare primarily as an antibacterial preservative agent in bacteriostatic saline. It has also been shown to have anesthetic properties, and has been demonstrated to cause less pain with infusion compared to lidocaine, while maintaining adequate pain relief. The use of bacteriostatic saline alone as an anesthetic for incisional procedures in the periocular area has not yet been studied. The purpose of this study was to determine whether bacteriostatic saline provides an adequate level of anesthesia for minor in-office eyelid procedures while allowing for reducing pain associated with medication infusion compared with traditional local anesthetic agents. To assess this, the investigators will recruit 150 patients aged 18 or older undergoing minor eyelid procedures including eyelid biopsies, chalazion removal from outpatient oculoplastics clinics at University of California, San Francisco. Patients will be randomized in a 1:1 fashion to undergo local anesthetic with either 1% lidocaine with 1:100,000 epinephrine or 0.9% bacteriostatic saline. Primary outcome measure will be pain level on a scale of 1-10 with regards to injection and procedure itself. These will be compared between the two groups. The investigators hypothesize that bacteriostatic saline is superior to lidocaine with epinephrine in terms of pain with injection, but will result in a similar pain level during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years old
2. Undergoing clinic-based periocular procedure

Exclusion Criteria:

1. Any other topical, oral or intravenous sedating medications given alongside procedure
2. Allergy to saline, lidocaine or epinephrine
3. Unable to provide consent due to cognitive impairment

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kersten, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California at San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson L, Martin S. Benzyl alcohol as an alternative local anesthetic. Ann Emerg Med. 1999 May;33(5):495-9. doi: 10.1016/s0196-0644(99)70335-5. PMID 10216324
- [Background] Minogue SC, Sun DA. Bacteriostatic saline containing benzyl alcohol decreases the pain associated with the injection of propofol. Anesth Analg. 2005 Mar;100(3):683-686. doi: 10.1213/01.ANE.0000148617.98716.EB. PMID 15728052
- [Background] Patterson P, Hussa AA, Fedele KA, Vegh GL, Hackman CM. Comparison of 4 analgesic agents for venipuncture. AANA J. 2000 Feb;68(1):43-51. PMID 10876451
- [Background] Miller L, Jensen MP, Stenchever MA. A double-blind randomized comparison of lidocaine and saline for cervical anesthesia. Obstet Gynecol. 1996 Apr;87(4):600-4. doi: 10.1016/0029-7844(95)00463-7. PMID 8602315
- [Background] Kruse RC, Kindle BJ, Wisniewski S, Presley J, Smith J, Sellon JL. Local Anesthesia Prior to Ultrasound-Guided Hip Joint Injections: A Double-Blind Randomized Controlled Trial of Bacteriostatic Saline versus Buffered Lidocaine. PM R. 2021 Aug;13(8):811-818. doi: 10.1002/pmrj.12489. Epub 2020 Nov 23. PMID 32935453
- [Background] Kwiat DM, Bersani TA, Bersani A. Increased patient comfort utilizing botulinum toxin type a reconstituted with preserved versus nonpreserved saline. Ophthalmic Plast Reconstr Surg. 2004 May;20(3):186-9. doi: 10.1097/01.iop.0000129012.09632.49. PMID 15167724
- [Background] Hunt SV, Malhotra R. Bacteriostatic preserved saline for pain-free periocular injections: review. Eye (Lond). 2022 Aug;36(8):1546-1552. doi: 10.1038/s41433-021-01925-z. Epub 2022 Jan 11. PMID 35017698
- [Background] Yuen VH, Dolman PJ. Comparison of three modified lidocaine solutions for use in eyelid anesthesia. Ophthalmic Plast Reconstr Surg. 1999 Mar;15(2):143-7. doi: 10.1097/00002341-199903000-00017. PMID 10189646
- [Background] Lugo-Janer G, Padial M, Sanchez JL. Less painful alternatives for local anesthesia. J Dermatol Surg Oncol. 1993 Mar;19(3):237-40. doi: 10.1111/j.1524-4725.1993.tb00342.x. PMID 8383150
- [Background] Oman KS, Fink R, Kleiner C, Makic MB, Wenger B, Hoffecker L, Mancuso M, Schmiege S, Cook P. Intradermal lidocaine or bacteriostatic normal saline to decrease pain before intravenous catheter insertion: a meta-analysis. J Perianesth Nurs. 2014 Oct;29(5):367-76. doi: 10.1016/j.jopan.2013.12.008. PMID 25261140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 95 patients with 110 lesions were recruited. There were 103 "encounters," creating duplicate patients in the two separate groups. The primary unit type analyzed was lesions. Participants had either 1, 2, or 3 lesions. Each lesion was randomized separately. Therefore, one participant could be part of both the bacteriostatic and lidocaine with epinephrine groups.
Units Other Than Participants: Lesions
Period: Overall Study
Arm/Group | Bacteriostatic Saline as Local Anesthesia | Lidocaine With Epinephrine as Local Anesthesia
Started | 55; 59 Lesions | 48; 51 Lesions
Completed | 55; 59 Lesions | 48; 51 Lesions
Not Completed | 0; 0 Lesions | 0; 0 Lesions

BASELINE CHARACTERISTICS:
Population: 95 patients with 110 lesions were recruited. There were 103 "encounters," creating duplicate patients in the two separate groups. The primary unit type analyzed was lesions. Participants had either 1, 2, or 3 lesions. Each lesion was randomized separately. Therefore, one participant could be part of both the bacteriostatic and lidocaine with epinephrine groups.
Units Other Than Participants: Lesions
Groups:
- Total: Total of all reporting groups
Arm/Group | Bacteriostatic Saline as Local Anesthesia | Lidocaine With Epinephrine as Local Anesthesia | Total
Number analyzed (Participants) | 55 | 48 | 95
Number analyzed (Lesions) | 59 | 51 | 110
Age, Continuous [Mean (Standard Deviation); unit: years]
  Baseline Population by Population | 58.5 (18.5) | 59.8 (16.2) | 59.1 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender Distribution: Female | 42 | 32 | 74
  Gender Distribution: Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Baseline Lesion Size [Mean (Standard Deviation); unit: Millimeters] | 3.2 (3.3) | 3.7 (3.7) | 3.5 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Pain on Injection
Description: Pain on a scale of 0-10 during injection process (0 being no pain, 10 being worst pain ever experienced). These will be patient-reported verbally and recorded immediately after injection.
Time Frame: 5 minutes
Population: Primary unit analyzed was lesions. Because each participant may have been randomized more than once, each participant may have more than one outcome. For this reason, outcome measures are expressed based on lesions rather than participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Lesions
Arm/Group | Bacteriostatic Saline as Local Anesthesia | Lidocaine With Epinephrine as Local Anesthesia
Number analyzed (Participants) | 55 | 48
Number analyzed (Lesions) | 59 | 51
score on a scale | 2.8 (2.4) | 3.6 (2.6)

2. Primary Outcome: Pain of Procedure
Description: Pain on a scale of 0-10 during procedure (0 being no pain, 10 being worst pain ever experienced). These will be patient-reported verbally and recorded immediately after procedure.
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Lesions
Arm/Group | Bacteriostatic Saline as Local Anesthesia | Lidocaine With Epinephrine as Local Anesthesia
Number analyzed (Participants) | 55 | 48
Number analyzed (Lesions) | 59 | 51
score on a scale | 4.9 (2.9) | 2.0 (2.7)

3. Secondary Outcome: Number of Lesions That Needed Additional Anesthesia to Complete Procedure
Description: Number of Lesions that Needed Additional Anesthesia to Complete Procedure
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Number; unit: lesions
Units Other Than Participants: Lesions
Arm/Group | Bacteriostatic Saline as Local Anesthesia | Lidocaine With Epinephrine as Local Anesthesia
Number analyzed (Participants) | 55 | 48
Number analyzed (Lesions) | 59 | 51
lesions | 33 | 5

4. Secondary Outcome: Bleeding Level
Description: Physician-assessed level of bleeding after procedure (mild, moderate, severe). These will be physician-reported verbally and recorded immediately after procedure.
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Number; unit: Number of lesions
Units Other Than Participants: Lesions
Arm/Group | Bacteriostatic Saline as Local Anesthesia | Lidocaine With Epinephrine as Local Anesthesia
Number analyzed (Participants) | 55 | 48
Number analyzed (Lesions) | 59 | 51
Number of lesions
  Number of Lesions with Mild Bleeding | 29 | 33
  Number of Lesions with Moderate Bleeding | 25 | 16
  Number of Lesions with Severe Bleeding | 4 | 0
  Number of Lesions with Unknown Bleeding Level | 1 | 2

ADVERSE EVENTS:
Time Frame: Monitored for approximately 10 minutes following injection
Description: At risk patients listed on patient, not procedure level
Arm/Group | Bacteriostatic Saline as Local Anesthesia | Lidocaine With Epinephrine as Local Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/48
Other Adverse Events (participants affected / at risk) | 0/55 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT05294640/Prot_SAP_002.pdf
  • Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT05294640/ICF_001.pdf